CLINICAL TRIAL: NCT04055285
Title: Effect of Renal Denervation on Atrial Fibrillation
Acronym: ERDAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor of Cardiology, School of Medicine, National and Kapodistrian University of Athens, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERDAF
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Arterial Hypertension; Atrial Fibrillation
Keywords: arterial hypertension; atrial fibrillation; renal denervation; autonomous nervous system; implantable loop recorder; continuous monitoring; burden; insertable cardiac monitor; resistant hypertension
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sympathetic Renal Denervation (Experimental): Sympathetic Renal Denervation
  Interventions: Procedure: Sympathetic Renal Denervation; Device: Implantable Loop Recorder
- Conventional treatment with drug therapy (Active Comparator): Conventional drug therapy of resistant hypertension
  Interventions: Device: Implantable Loop Recorder

INTERVENTIONS:
Procedure: Sympathetic Renal Denervation — Catheter-based sympathetic renal denervation (RDN) using radiofrequency, ultrasound, or perivascular injection of neurotoxic agents such as alcohol has been introduced as a minimally invasive alternative treatment option for patients with resistant hypertension. RDN consists of endovascular catalysis of the kidney sympathetic nerves running in the wall of the renal arteries.
  Arms: Sympathetic Renal Denervation
Device: Implantable Loop Recorder — Implantable Loop Recorders (ILRs) are small, subcutaneously implanted devices that are able to detect and store atrial fibrillation episodes lasting longer than 2 minutes with high sensitivity (96.1-100%) and good specificity (67-85.4%) for a period of up to three years.
  Other Names: Insertable Cardiac Monitor

SUMMARY:
The purpose of the ERDAF study (Effect of Renal Denervation on Atrial Fibrillation) is to evaluate the renal sympathetic denervation in patients with resistant arterial hypertension and symptomatic paroxysmal or persistent atrial fibrillation(AF) in order to show if there is a reduction in the AF-related symptoms, the AF recurrence rate, and the total burden (symptomatic and/or asymptomatic) of the arrhythmia. To the best of our knowledge, ERDAF is the first randomized study, which is going to evaluate the effect of RDN [without pulmonary vein isolation (PVI)] on AF recurrence profile and AF ''burden'' using continuous long-term rhythm monitoring via ILRs for a period of 18 months.

Hypothesis

Renal sympathetic denervation in patients with resistant hypertension and symptomatic paroxysmal or persistent atrial fibrillation reduces AF recurrences, total AF "burden" (asymptomatic / symptomatic) and limits the AF-related symptoms.

DETAILED DESCRIPTION:
In arterial hypertension (AH), a significant proportion of patients, despite the optimal medical therapy, do not achieve adequate blood pressure (BP) control (resistant hypertension). Renal sympathetic denervation (RDN) is a novel alternative minimally invasive therapeutic option for patients with resistant AH. Recent data has shown that RDN with or without pulmonary vein isolation (PVI) may also have a positive impact on the management of patients with paroxysmal or persistent atrial fibrillation (AF). However, there is no randomized study, to date, suggesting that RDN itself (without PVI) reduces the AF recurrences, symptoms, and the total burden of the arrhythmia. The purpose of this study [Effect of Renal Denervation on Atrial Fibrillation (ERDAF)] is to evaluate the RDN (without PVI) in patients with resistant AH and symptomatic paroxysmal or persistent AF in order to show if there is benefit in the incidence of AF recurrences, the total AF burden (symptomatic and asymptomatic) as well as the BP control. This is a single-center, randomized study in which thirty (30) patients with resistant AH and symptomatic paroxysmal or persistent AF will be randomized (1:1) after sinus rhythm restoration and implantation of an implantable loop recorder (ILR), in either RDN (n=15) or conventional treatment of resistant AH with optimal drug therapy (n=15). Patients will be followed-up every three months and for a period of 18 months after the implantation of the ILR. The first three months after RDN will be excluded from our final analysis (blanking period). The primary endpoint will be the change in the total AF burden (Total time in AF during the follow-up period). Secondary endpoints will include the change in the symptomatic and asymptomatic burden of AF, the time to detect the first AF recurrence (symptomatic and/or asymptomatic)-early recurrence of AF after RDN, and the change in BP during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Patients >18 years with resistant hypertension [Systolic Blood Pressure (SBP) ≥ 140 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 90 mmHg despite treatment with ≥ 3 antihypertensive drugs of various classes, including a diuretic) and symptomatic paroxysmal or persistent AF will be included in the study after sinus rhythm restoration

Exclusion Criteria:

1. Patients with permanent AF or patients with long-standing persistent AF as defined by the current ESC guidelines for the management of AF1.
2. Patients with a glomerular filtration rate (eGFR)] <45 ml / min / 1.73 m2 calculated using the CKD-EPI43.
3. Patients with secondary arterial hypertension.
4. Patients with an established diagnosis of resistant hypertension <6 months.
5. Patients with severe renal artery stenosis or previous renal artery angioplasty.
6. Patients who have undergone or are about to undergo pulmonary vein isolation.
7. Patients with left end-diastolic ventricle diameter >60 mm in men or >55mm in women.
8. Patients with a left ventricular ejection fraction <35% in the transthoracic echocardiogram (TTE).
9. Patients with AF possible reversible causes (pulmonary embolism, acute coronary syndromes, thyrotoxicosis, alcohol abuse, etc.)
10. Patients with heart failure in NYHA III-IV stage.
11. Patients with life expectancy <1 year.
12. Pregnant women.
13. Patients who are unable to give consent to participate in the study.
14. Patients who do not wish to give written consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in the total AF "burden" (symptomatic and asymptomatic AF burden) during the follow-up period. | From 3 months to 18 months.The first three months after RDN will be excluded from our final analysis (blanking period)
  AF "burden": The amount of time (minutes or hours) the patient is in AF out of the total follow-up period.

SECONDARY OUTCOMES:
Change in the symptomatic AF "burden" during the follow-up period. | From 3 months to 18 month.The first three months after RDN will be excluded from our final analysis (blanking period)
  Symptomatic AF ''burden'': The amount of time (minutes or hours) in which the patient is in AF, perceived by the patient AF, out of the total follow-up period.
Change in asymptomatic AF "burden" during the follow-up period. | From 3 months to 18 months. The first three months after RDN will be excluded from our final analysis (blanking period)
  Asymptomatic AF "burden": The amount of time (minutes or hours) in which the patient is in AF that the patient does not perceive out of the total follow-up period.
The time interval for the detection of the first AF recurrence after the ILR implantation during the follow-up period. | From 3 months to 18 months. The first three months after RDN will be excluded from our final analysis (blanking period)
The time interval for detection of the first symptomatic recurrence of the arrhythmia after the ILR implantation during the follow-up period. | From 3 months to 18 months. The first three months after RDN will be excluded from our final analysis (blanking period)
Change in blood pressure (systolic, diastolic, and mean blood pressure) as measured by 24-hour ambulatory blood pressure monitoring (ABPM) during the follow-up period. | From 3 months to 18 months. The first three months after RDN will be excluded from our final analysis (blanking period)
Change in office blood pressure (systolic, diastolic). | From 3 months to 18 months. The first three months after RDN will be excluded from our final analysis (blanking period)

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos P Tsioufis, MD, PhD, Study Director — First Cardiology Deparment, Hippokration Hospital, Athens, Greece; Panteleimon E Papakonstantinou, MD, PhD, Principal Investigator — First Cardiology Deparment, Hippokration Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Europace. 2016 Nov;18(11):1609-1678. doi: 10.1093/europace/euw295. Epub 2016 Aug 27. No abstract available. PMID 27567465
- [Background] Zoni-Berisso M, Lercari F, Carazza T, Domenicucci S. Epidemiology of atrial fibrillation: European perspective. Clin Epidemiol. 2014 Jun 16;6:213-20. doi: 10.2147/CLEP.S47385. eCollection 2014. PMID 24966695
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Tsioufis C, Ziakas A, Dimitriadis K, Davlouros P, Marketou M, Kasiakogias A, Thomopoulos C, Petroglou D, Tsiachris D, Doumas M, Skalidis E, Karvounis C, Alexopoulos D, Vardas P, Kallikazaros I, Stefanadis C, Papademetriou V, Tousoulis D. Blood pressure response to catheter-based renal sympathetic denervation in severe resistant hypertension: data from the Greek Renal Denervation Registry. Clin Res Cardiol. 2017 May;106(5):322-330. doi: 10.1007/s00392-016-1056-z. Epub 2016 Dec 12. PMID 27957627
- [Background] Grassi G, Mark A, Esler M. The sympathetic nervous system alterations in human hypertension. Circ Res. 2015 Mar 13;116(6):976-90. doi: 10.1161/CIRCRESAHA.116.303604. PMID 25767284
- [Background] Tsioufis C, Dimitriadis K, Kasiakogias A, Kalos T, Liatakis I, Koutra E, Nikolopoulou L, Kordalis A, Ella RO, Lau EO, Grassi G, Papademetriou V, Tousoulis D. Effects of multielectrode renal denervation on elevated sympathetic nerve activity and insulin resistance in metabolic syndrome. J Hypertens. 2017 May;35(5):1100-1108. doi: 10.1097/HJH.0000000000001262. PMID 28106665
- [Background] Simantirakis EN, Papakonstantinou PE, Chlouverakis GI, Kanoupakis EM, Mavrakis HE, Kallergis EM, Arkolaki EG, Vardas PE. Asymptomatic versus symptomatic episodes in patients with paroxysmal atrial fibrillation via long-term monitoring with implantable loop recorders. Int J Cardiol. 2017 Mar 15;231:125-130. doi: 10.1016/j.ijcard.2016.12.025. Epub 2016 Dec 21. PMID 28041713
- [Background] Bettoni M, Zimmermann M. Autonomic tone variations before the onset of paroxysmal atrial fibrillation. Circulation. 2002 Jun 11;105(23):2753-9. doi: 10.1161/01.cir.0000018443.44005.d8. PMID 12057990
- [Background] Lombardi F, Tarricone D, Tundo F, Colombo F, Belletti S, Fiorentini C. Autonomic nervous system and paroxysmal atrial fibrillation: a study based on the analysis of RR interval changes before, during and after paroxysmal atrial fibrillation. Eur Heart J. 2004 Jul;25(14):1242-8. doi: 10.1016/j.ehj.2004.05.016. PMID 15246643
- [Background] Papademetriou V, Doumas M, Tsioufis K. Renal Sympathetic Denervation for the Treatment of Difficult-to-Control or Resistant Hypertension. Int J Hypertens. 2011;2011:196518. doi: 10.4061/2011/196518. Epub 2011 Mar 30. PMID 21629864
- [Background] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Baranova V, Turov A, Shirokova N, Karaskov A, Mittal S, Steinberg JS. A randomized comparison of pulmonary vein isolation with versus without concomitant renal artery denervation in patients with refractory symptomatic atrial fibrillation and resistant hypertension. J Am Coll Cardiol. 2012 Sep 25;60(13):1163-70. doi: 10.1016/j.jacc.2012.05.036. Epub 2012 Sep 5. PMID 22958958
- [Background] Vollmann D, Sossalla S, Schroeter MR, Zabel M. Renal artery ablation instead of pulmonary vein ablation in a hypertensive patient with symptomatic, drug-resistant, persistent atrial fibrillation. Clin Res Cardiol. 2013 Apr;102(4):315-8. doi: 10.1007/s00392-012-0529-y. Epub 2012 Dec 14. No abstract available. PMID 23239408
- [Background] Qiu M, Yin Y, Shan Q. Renal sympathetic denervation versus antiarrhythmic drugs for drug-resistant hypertension and symptomatic atrial fibrillation (RSDforAF) trial: study protocol for a randomized controlled trial. Trials. 2013 Jun 11;14:168. doi: 10.1186/1745-6215-14-168. PMID 23759000
- [Background] Feyz L, Theuns DA, Bhagwandien R, Strachinaru M, Kardys I, Van Mieghem NM, Daemen J. Atrial fibrillation reduction by renal sympathetic denervation: 12 months' results of the AFFORD study. Clin Res Cardiol. 2019 Jun;108(6):634-642. doi: 10.1007/s00392-018-1391-3. Epub 2018 Nov 10. PMID 30413869
- [Background] Kosiuk Md J, Pokushalov Md Phd E, Hilbert Md S, Hindricks Md G, Bollmann Md PhD A, S Steinberg Md J. The Role of Renal Sympathetic Denervation in Atrial Fibrillation. J Atr Fibrillation. 2014 Feb 28;6(5):987. doi: 10.4022/jafib.987. eCollection 2014 Feb-Mar. PMID 27957040
- [Background] Charitos EI, Ziegler PD, Stierle U, Robinson DR, Graf B, Sievers HH, Hanke T. Atrial fibrillation burden estimates derived from intermittent rhythm monitoring are unreliable estimates of the true atrial fibrillation burden. Pacing Clin Electrophysiol. 2014 Sep;37(9):1210-8. doi: 10.1111/pace.12389. Epub 2014 Mar 25. PMID 24665972
- [Background] Simantirakis EN, Papakonstantinou PE, Kanoupakis E, Chlouverakis GI, Tzeis S, Vardas PE. Recurrence rate of atrial fibrillation after the first clinical episode: A prospective evaluation using continuous cardiac rhythm monitoring. Clin Cardiol. 2018 May;41(5):594-600. doi: 10.1002/clc.22904. Epub 2018 May 14. PMID 29761516
- [Background] Papakonstantinou PE, Simantirakis EN. Long-term rhythm monitoring with an implantable loop recorder in patients after the first clinical atrial fibrillation episode. Towards an individualized management. Minerva Cardioangiol. 2019 Apr;67(2):121-130. doi: 10.23736/S0026-4725.19.04883-7. Epub 2019 Feb 5. PMID 30724269
- [Background] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169
- [Background] Ciconte G, Saviano M, Giannelli L, Calovic Z, Baldi M, Ciaccio C, Cuko A, Vitale R, Giacopelli D, Conti M, Lipartiti F, Giordano F, Maresca F, Moscatiello M, Vicedomini G, Santinelli V, Pappone C. Atrial fibrillation detection using a novel three-vector cardiac implantable monitor: the atrial fibrillation detect study. Europace. 2017 Jul 1;19(7):1101-1108. doi: 10.1093/europace/euw181. PMID 27702865